CLINICAL TRIAL: NCT02071537
Title: A Phase 1 Study of Chloroquine in Combination With Carboplatin/Gemcitabine in Advanced Solid Tumors
Brief Title: Chloroquine in Combination With Carboplatin/Gemcitabine in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-EXP-13-01
Record Dates: First submitted 2014-02-19; First posted 2014-02-26 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Malignant Neoplasm; Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Chloroquine; chloroquine diphosphate; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chloroquine with Carboplatin/Gemcitabine (Experimental): Chloroquine administered orally daily to start one week prior to Carboplatin (AUC5)/Gemcitabine (1250mg/m2). Chloroquine dose is escalating.
  Interventions: Drug: Chloroquine; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Chloroquine — Dose is 50, 100, 150, and 200 mg per day cohorts. It is given one week prior to the initiation of chemotherapy and then given for four 21 day cycles in combination with chemotherapy.
  Other Names: Chloroquine Phosphate; Aralen
Drug: Carboplatin — Administered day 1 of each 21 day cycle for 4-6 cycles.
  Other Names: Paraplatin; CBDCA
Drug: Gemcitabine — Administered days 1 and 8 of each 21 day cycle for 4-6 cycles.
  Other Names: Gemzar

SUMMARY:
The purpose of this research study is to test the safety of chloroquine in combination with carboplatin and gemcitabine and see what effects (good and bad) it has on advanced solid tumors.

Also, the research study will be increasing the dose of chloroquine to find the highest dose of chloroquine that can be given in combination with carboplatin and gemcitabine without causing severe side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a malignancy that is metastatic or unresectable and for which either standard curative measures do not exist or are no longer effective and carboplatin/gemcitabine is considered a reasonable treatment option whether first line or acceptable and approved combination therapy.
* Age >18 years of age.
* Performance status less than or equal 2 (Karnofsky >60%)
* Life expectancy of greater than 3 months.
* Adequate labs
* Measurable disease

Exclusion Criteria:

* Current treatment with any other investigational agents.
* Patients with untreated brain metastases
* History of allergic reaction attributed to compounds of similar chemical or biologic composition to chloroquine or other agents used in study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05-13 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of chloroquine when combined with Carboplatin/Gemcitabine | Up to 12 months

SECONDARY OUTCOMES:
Time to Disease Progression | Up to 24 months
Time of Overall Survival | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nagla Abdel-Karim, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Cancer Institute, Cincinnati, Ohio, United States